CLINICAL TRIAL: NCT03571100
Title: Patient Comfort and Antimicrobial Efficacy With Aqueous Chlorhexidine Versus Povidine-Iodine (Betadine) as Ocular Surface Disinfectant Prior to Intravitreal Injection
Brief Title: Comfort and Antimicrobial Efficacy of Chlorhexidine vs Betadine for Intravitreal Injections
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MidAtlantic Retina (Other)
Responsible Party: Sponsor-Investigator, MidAtlantic Retina, Dr Sunir Garg MD, Wills Eye
Organization: Wills Eye (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-692E
Record Dates: First submitted 2018-05-10; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Age-related Macular Degeneration; Diabetic Vascular Diseases; Proliferative Retinopathy; Retina Vein Occlusion
MeSH Terms: conditions — Macular Degeneration; Diabetic Angiopathies | interventions — Chlorhexidine; Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Randomized prospective trial
Who Masked: Participant
Masking Description: The participant will be masked to which drug they receive, the investigator performing the analysis will also be masked
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Povidine-Iodine (Active Comparator): Bilateral injections patients receiving Povidine-Iodine in right eye, chlorhexidine in the left eye
  Interventions: Drug: Povidine-Iodine
- Chlorhexidine (Active Comparator): Bilateral injections patients receiving Povidine-Iodine in left eye, chlorhexidine in the right eye
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Chlorhexidine — Chlorhexidine administration prior to intravitreal injection (compared to gold standard povidine-iodine)
  Other Names: Aqueous chlorhexidine
  Arms: Chlorhexidine
Drug: Povidine-Iodine — Povidine iodine administration prior to intravitreal injection (compared to chlorhexidine)
  Other Names: Betadine
  Arms: Povidine-Iodine

SUMMARY:
The purpose of this prospective interventional study is to compare patient experience, ocular surface irritation, and bacterial colony counts and microbial spectrum between povidine iodine and aqueous chlorhexidine as ocular surface antiseptic prior to intravitreal injection

DETAILED DESCRIPTION:
This is a single center prospective study comparing antiseptic efficacy and ocular surface irritation with PI (povidine iodine) and AC (aqueous chlorhexidine). Patients will be recruited in the clinical offices of the Retina Service of Wills and Hospital/Mid Atlantic Retina clinic offices. Patients who are determined to require bilateral intravitreal injections of an anti-VEGF (vascular endothelial growth factor) agents by a retina specialist at their regularly scheduled retina appointment will be evaluated for qualification by study personnel. Patients who meet inclusion criteria will be identified and informed consent will be obtained. Prior to injection, topical anesthetic (0.5% proparacaine, Alcon) will be instilled in both eyes. Study personnel will obtain four samples from the superior and inferior fornices of the upper and lower lids of both eyes using swabs (COPAN ESwab, ThermoFisher Scientific) for patients enrolled at Wills. Topical antisepsis will then be applied, the first eye will be randomized to one drop of either PI 5% or AC 0.1% and the second eye will receive the other agent. One minute after instillation of the eye drop to each eye, patients will rate their pain in each eye using the Wong-Baker (smiley face) rating scale. The injections will then be performed by the treating retina specialist. Following the injection, a second conjunctival culture will be taken in an identical manner to the first for patients enrolled at Wills. Study personnel will then instill fluorescein dye (fluorescein sodium ophthalmic, BioGlo) into each eye, and a brief slit lamp examination will be performed. Study personnel will record surface findings according to the Ocular Surface Score and a numerical score for each eye will be determined. On post-injection day one study personnel will call the patient and ask to rate the pain in each eye using the same verbal numerical rating scale. No additional clinic visits will be required as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Current patient of the Wills Eye Hospital Retina Service including all Mid Atlantic Retina offices
* Clinical indication of bilateral intravitreal injection as determined by the treating retina specialist for a diagnosis of age-related macular degeneration, diabetic macular edema, proliferative retinopathy or macular edema associated with retina vein occlusion.
* Age greater than 18.

Exclusion Criteria:

* Documented allergy to PI or AC
* Current diagnosis of infectious keratitis
* History of unilateral contact lens wear in the past 30 days
* Current unilateral use of prescription eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-05-06 (Estimated); Study Completion 2019-05-06 (Estimated)

PRIMARY OUTCOMES:
Patient Comfort | One day following injection
  Patient Comfort using the Wong Baker FACES Pain Scale [Scale: 0(No pain) - 10 (Worst Pain)]

SECONDARY OUTCOMES:
Culture of conjunctiva for bacteria | 7 days
  Microbial flora
Patient Comfort | I minute after drop instilled
  Patient Comfort using the Wong Baker FACES Pain Scale [Scale: 0(No pain) - 10 (Worst Pain)]

CONTACTS AND LOCATIONS:
Overall Officials: Sunir Garg, MD, Principal Investigator — MidAtlantic Retina
Locations (1):
- MidAtlantic Retina, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali FS, Jenkins TL, Boparai RS, Obeid A, Ryan ME, Wibblesman TD, Chiang A, Garg SJ; Post-Injection Endophthalmitis Study Group. Aqueous Chlorhexidine Compared with Povidone-Iodine as Ocular Antisepsis before Intravitreal Injection: A Randomized Clinical Trial. Ophthalmol Retina. 2021 Aug;5(8):788-796. doi: 10.1016/j.oret.2020.11.008. Epub 2020 Nov 20. PMID 33221515